CLINICAL TRIAL: NCT03577509
Title: Pharmacokinetics, Safety and Tolerability of Single Infusion of Amphotericin B Colloidal Dispersion In Healthy Subjects in China
Brief Title: Single Dose Escalations Study of Amphotericin B Colloidal Dispersion In Healthy Subjects in China
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LXMSB201701/PRO
Record Dates: First submitted 2018-05-28; First posted 2018-07-05 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-05

CONDITIONS: Invasive Fungal Disease
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABCD (Experimental): Group1: 0.5mg/kg Group2: 1.0mg/kg Group3: 1.5mg/kg
  Interventions: Drug: ABCD

INTERVENTIONS:
Drug: ABCD — Intravenous infusion of dexamethasone 5mg before ABCD intravenous administration; Single infusion.

SUMMARY:
The purpose of this trial is to evaluate the pharmacokinetics of single intravenous of Amphotericin B Colloidal Dispersion(ABCD)in Chinese healthy subjects.

DETAILED DESCRIPTION:
Primary Objective: Evaluation the pharmacokinetics, safety and tolerability of single intravenous of ABCD in Chinese healthy subjects.

Secondary Objective: Evaluation the safety and tolerability of single intravenous of ABCD in Chinese healthy subjects.

Exploratory Objective:Evaluation the effect of single intravenous ABCD on early renal injury indicators (KIM-1 and cystatin C) in Chinese healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 19 to 26 kg/m2, inclusive 19 and 26. BMI = weight (kg)/[height(m)]2.
* Subjects are fully informed and voluntarily consent to participate in this study.

Exclusion Criteria:

* History of allergy or hypersensitivity.
* Presence of any acute or chronic medical condition within 3 months prior to investigational products administration, including but not limited to: hepatic, gastrointestinal, renal, hematologic (including coagulation), pulmonary, neurologic, respiratory, endocrine, or cardiovascular system abnormalities; psychiatrical disease including major psychiatric disorders (e.g., schizophrenia, bipolar disorder); acute infection; or other conditions that would interfere with the absorption, distribution, metabolism, or excretion of drugs.
* During the screening period, abnormal and clinically significant of physical examination, vital signs, laboratory examination, etc.
* A positive result in hepatitis B surface antigen (HBsAg), hepatitis B e antigen (HBeAg), anti-hepatitis C virus (HCV) antibodies, a syphilis test, or an human immunodeficiency virus (HIV) test.
* Lost blood or donated more than 400 mL of blood within 3 months prior to the screening.
* Participation in a clinical drug study 30 days prior to present study.
* Use of any other drugs within 2 weeks prior to the screening.
* Subjects planning to give birth or donate sperm during the study or within 3 months after the study.
* The partner of the subject is unwilling to take effective contraceptive measures.
* Other unfavorable factors diagnosed by investigators.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of single infusion of ABCD | before infusion and at the midpoint and end of the infusion;and at 15 and 30 min;1,2,4,7,10,24,48,72,120,168,240,336,408,504,576 and 672hour postinfusion
  Peak Plasma Concentration,.
Pharmacokinetics of single infusion of ABCD | before infusion and at the midpoint and end of the infusion;and at 15 and 30 min;1,2,4,7,10,24,48,72,120,168,240,336,408,504,576 and 672hour postinfusion
  Area under the plasma concentration versus time curve

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zhang, Ph.D, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang ZW, Yu JC, Wang JJ, Chen YC, Wu JF, Chen YJ, Cao GY, Yang HJ, He JJ, Dai JY, Zhang JY, Zhang W, Yuan J, Li CL, Xu FY, Wang K, Wu XJ, Zhang J. Pharmacokinetics and Safety of Single-Dose Amphotericin B Colloidal Dispersion in Healthy Chinese Subjects and Population Pharmacokinetic/Pharmacodynamic Analysis to Inform Clinical Efficacy in Invasive Infections Caused by Candida albicans. Clin Ther. 2021 Nov;43(11):1921-1933.e7. doi: 10.1016/j.clinthera.2021.09.012. Epub 2021 Oct 20. PMID 34686365